CLINICAL TRIAL: NCT05502640
Title: The Effect of Chicken Model in Teaching Episiotomy Repair on Satisfaction, Self-Confidence, and Anxiety Levels of Midwifery Students
Brief Title: Chicken Model in Teaching Episiotomy Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, İlknur Münevver Gönenç, Associate Professor Dr., Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 289
Record Dates: First submitted 2022-04-25; First posted 2022-08-16 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Episiotomy Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sponge group (Other): Control group
  Interventions: Other: Routine Education model
- Chicken group (Experimental)
  Interventions: Other: Education model

INTERVENTIONS:
Other: Education model — Chicken legs will be used for each student in the study. Intermittent and continuous suture techniques will be studied on the incision made on the chicken leg.
  Arms: Chicken group
Other: Routine Education model — In the study, 15 cm x 20 cm sponge will be used for each student. Intermittent and continuous suture techniques will be practiced on the sponge.
  Other Names: Sponge Group
  Arms: sponge group

SUMMARY:
The aim of this study is to determine the effect of chicken use in episiotomy repair training of midwifery students on students' satisfaction, self-confidence and anxiety levels.

Hypotheses H01 There is no difference between the satisfaction score of the chicken group and the satisfaction score of the control group in episiotomy repair training.

H02 In episiotomy repair training, there is no difference between the self-confidence score of the chicken group and the self-confidence score of the control group.

H03 There is no difference between the anxiety score of the chicken group and the anxiety score of the control group in episiotomy repair training.

ELIGIBILITY:
Inclusion Criteria:

* Midwifery students who were registered in the midwifery department in the 2020-2021 academic year and take childbearing course,
* Students over the age of 18

Exclusion Criteria:

* Having previously received training on episiotomy and its repair,
* Students who fill in the data collection forms incompletely will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in The State-Trait Anxiety Inventory (STAI) | immediately before the training, immediately after the training and immediately after the clinical practice.
  The inventory was developed by Spielberger et al. in 1970. An adaptation, validity, and reliability study of the State-Trait Anxiety Scale in Turkish was conducted by Oner and Le Compte in 1983. The scale consists of two subdimensions: the state anxiety has 20 items and is used to determine what is felt at a specific moment under certain conditions, and the trait anxiety has 20 items and is used to determine what has been felt in the last 7 days. High scores from each subscale indicate a high level of anxiety.
  STAI-S consist of 20 items with four points Likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Change in satisfaction | immediately before the training, immediately after the training and immediately after the clinical practice.
  Visual Analog Scale is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfaction and a score of 0 pointed to no satisfaction.
Self-Sufficiency | immediately before the training, immediately after the training and immediately after the clinical practice.
  Visual Analog Scale (VAS)- assessed by adequate vision. For each item, students rated their sense of self-sufficiency on a scale of 0 (very inadequate) to 10 (very adequate).
The Student Satisfaction and Self-Confidence in Learning Scale | immediately after training
  This instrument is a 13-item scale used to measure student satisfaction with the simulation activity (5 items) and self-confidence in learning (8 items). Responses are rated on a 5-point Likert scale with values ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher satisfaction and greater levels of self confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided